CLINICAL TRIAL: NCT02788123
Title: Phase IV, Multicenter, Open Label, Randomized Study in Parallel Groups To Assess The Efficacy And Safety Of Bismuth Tripotassium Dicitrate (De-Nol®) In Combination With Pantoprazole And Pantoprazole Monotherapy In Treatment Of Patients With NSAID Induced Gastropathy
Brief Title: A Study To Assess The Efficacy And Safety Of Bismuth Tripotassium Dicitrate (De-Nol) In Combination With Pantoprazole And Pantoprazole Monotherapy In Treatment Of Subjects With Nonsteroidal Anti-Inflammatory Drugs (NSAID)-Induced Gastropathy
Acronym: BiGARD
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Internal reassessment of the medicinal product development strategy by Sponsor
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3593-MA-3026-RU
Record Dates: First submitted 2016-05-27; First posted 2016-06-02 (Estimated); Last update posted 2017-09-21 (Actual); Status verified 2017-09

CONDITIONS: NSAID-induced Gastropathy
Keywords: De-Nol; NSAID-induced gastropathy; Pantoprazole; Bismuth tripotassium dicitrate; Russia
MeSH Terms: interventions — bismuth tripotassium dicitrate; Pantoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bismuth tripotassium dicitrate and pantoprazole (Experimental): Participants will receive bismuth tripotassium dicitrate (twice daily) and pantoprazole (once daily) as single tablets
  Interventions: Drug: bismuth tripotassium dicitrate; Drug: pantoprazole
- pantoprazole (Active Comparator): Participants will receive pantoprazole (once daily) as single tablet
  Interventions: Drug: pantoprazole

INTERVENTIONS:
Drug: bismuth tripotassium dicitrate — oral
  Other Names: De-Nol
  Arms: bismuth tripotassium dicitrate and pantoprazole
Drug: pantoprazole — oral
  Other Names: Controloc

SUMMARY:
The main purpose of this study is to evaluate clinical efficacy of bismuth tripotassium dicitrate (De-Nol) in combination with pantoprazole versus pantoprazole monotherapy in subjects with NSAID-induced gastropathy in 14±2 days of treatment.

DETAILED DESCRIPTION:
This study has a screening period (up to 3±2 days duration). Randomization will be held in each stratum (H. pylori-positive and H. pylori-negative) on the Visit 1. Treatment period will consist of 2 visits: Visit 2 (up to 14±2 days after Visit 1) in subjects with completely healed ulcer(s) and erosions after control esophagogastroduodenoscopy (EGDS) and Visit 3 (up to 28±2 days after Visit 1) in subjects with not healed ulcers and erosions after control EGDS on Visit 2. The period of follow-up safety assessments will last 1 week after the end of the study treatment

ELIGIBILITY:
Inclusion Criteria:

* Verified diagnosis of NSAID-induced gastropathy:

  * Presence of gastric ulcer(s) and/or erosions (modified Lanza score greater than or equal to 5) based on EGDS findings at screening and;
  * NSAIDs administration within 7 days before screening.
* Negative pregnancy test at screening and at Visit 1 (for females only using test strip to detect chorionic gonadotropin in urine),
* Subjects' consent to use a reliable contraception method starting from screening throughout the whole study and for 1 week after its termination.

Exclusion Criteria:

* Severe complications of NSAID-gastropathy (bleedings, perforations, etc.)
* The subjects requiring concomitant therapy using the drugs specified in "Forbidden concomitant therapy".
* Ulcerative esophagitis grade C and higher according to Los-Angeles classification.
* Expressed hepatic and renal impairment.
* Any esophageal and gastric surgery that can make subject ineligible for study participation.
* Abuse of psychoactive substances including alcohol which may interfere with the subject's participation and fulfillment of all the protocol requirements.
* Participation in other clinical studies within 30 days prior to Screening Visit.
* Administration of bismuth products less than 2 months prior to screening.
* Administration of PPIs or histamine Н2-receptor antagonists less than 2 weeks prior to screening.
* Hypersensitivity to any of the components of the study drugs or contraindications to them.
* Pregnancy and lactation.
* Inability to perform follow-up EGDS after 2 and/or 4 weeks of the study.
* Any condition or concomitant disease and laboratory parameter abnormalities which renders the subject ineligible for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2017-05-29 (Actual); Study Completion 2017-06-13 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects in each group reaching complete healing of NSAID-induced gastropathy at week 2 of therapy | Week 2
  Modified Lanza score 0-2 (inclusively) shall be considered as healing. The modified Lanza scale is utilized to grade the degree of gastritis

SECONDARY OUTCOMES:
Proportion of subjects reaching complete healing of NSAID-induced gastropathy in H.pylori-negative subjects in each treatment group at week 2 | Week 2
  Modified Lanza scale 0-2 scores (inclusively) shall be considered as complete healing
Proportion of subjects reaching complete healing of NSAID-induced gastropathy in H.pylori-positive subjects in each treatment group at week 2 | Week 2
  Modified Lanza scale 0-2 scores (inclusively) shall be considered as complete healing
Proportion of subjects reaching complete healing of NSAID-induced gastropathy in H.pylori-negative subjects in each treatment group at week 4 | Week 4
  Subjects reached complete healing of NSAID-induced gastric ulcers and erosions by Visit 2 shall also be analyzed
Proportion of subjects reaching complete healing of NSAID-induced gastropathy in H.pylori-positive subjects in each treatment group at week 4 | Week 4
  Subjects reached complete healing of NSAID-induced gastric ulcers and erosions by Visit 2 shall also be analyzed
Proportion of subjects reaching complete healing of NSAID-induced gastropathy in subjects with NSAID-induced gastropathy with modified Lanza scale greater than or equal to 5 and <7 at screening in each treatment group at week 2 | Week 2
  The modified Lanza scale is utilized to grade the degree of gastritis. Modified Lanza scale 0-2 scores (inclusively) shall be considered as complete healing
Proportion of subjects reaching complete healing of NSAID-induced gastropathy in subjects with NSAID-induced gastropathy with modified Lanza scale =7 at screening in each treatment group at week 2 | Week 2
  The modified Lanza scale is utilized to grade the degree of gastritis. Modified Lanza scale 0-2 scores (inclusively) shall be considered as complete healing
Proportion of subjects reaching complete healing of NSAID-induced gastropathy in subjects with NSAID-induced gastropathy with modified Lanza scale greater than or equal to 5 and <7 at screening in each treatment group at week 4 | Week 4
  The modified Lanza scale is utilized to grade the degree of gastritis. Modified Lanza scale 0-2 scores (inclusively) shall be considered as complete healing. Subjects reached complete healing of NSAID-induced gastric ulcers and erosions by Visit 2 shall also be analyzed
Proportion of subjects reaching complete healing of NSAID-induced gastropathy in subjects with NSAID-induced gastropathy with modified Lanza scale =7 at screening in each treatment group at week 4 | Week 4
  The modified Lanza scale is utilized to grade the degree of gastritis. Modified Lanza scale 0-2 scores (inclusively) shall be considered as complete healing. Subjects reached complete healing of NSAID-induced gastric ulcers and erosions by Visit 2 shall also be analyzed
Proportion of subjects reaching complete healing of NSAID-induced gastropathy in each treatment group at week 4 | Week 4
  Subjects reached complete healing of NSAID-induced gastric ulcers and erosions by Visit 2 shall also be analyzed
Changes in modified Lanza as compared to visit 1 (baseline) in H.pylori-negative subjects in each treatment group | Baseline, week 2 and week 4
  The modified Lanza scale is utilized to grade the degree of gastritis
Changes in modified Lanza as compared to visit 1 (baseline) in H.pylori-positive subjects in each treatment group | Baseline, week 2 and week 4
  The modified Lanza scale is utilized to grade the degree of gastritis
Changes in modified Lanza as compared to Visit 1 (baseline) in subjects with NSAID-induced gastropathy with modified Lanza scale greater than or equal to 5 and <7 at screening in each treatment group | Baseline, week 2 and week 4
  The modified Lanza scale is utilized to grade the degree of gastritis
Changes in modified Lanza as compared to Visit 1 (baseline) in subjects with NSAID-induced gastropathy with modified Lanza scale =7 at screening in each treatment group | Baseline, week 2 and week 4
  The modified Lanza scale is utilized to grade the degree of gastritis
Changes in modified Lanza as compared to visit 1 (baseline) in each treatment group | Baseline, week 2 and week 4
  The modified Lanza scale is utilized to grade the degree of gastritis
Changes in GSRS as compared to visit 1 (baseline) in H.pylori-negative subjects in each treatment group | Baseline, week 2 and week 4
  Gastrointestinal Symptom Rating Scale (GSRS). The GSRS contains a list of questions on subject's well-being within the period from subject's last visit to study site
Changes in GSRS as compared to visit 1 (baseline) in H.pylori-positive subjects in each treatment group | Baseline, week 2 and week 4
  Gastrointestinal Symptom Rating Scale (GSRS). The GSRS contains a list of questions on subject's well-being within the period from subject's last visit to study site
Changes in GSRS as compared to Visit 1 (baseline) in subjects with NSAID-induced gastropathy with modified Lanza scale greater than or equal to 5 and <7 at screening in each treatment group | Baseline, week 2 and week 4
  The GSRS contains a list of questions on subject's well-being within the period from subject's last visit to study site. The modified Lanza scale is utilized to grade the degree of gastritis
Changes in GSRS as compared to Visit 1 (baseline) in subjects with NSAID-induced gastropathy with modified Lanza scale =7 at screening in each treatment group | Baseline, week 2 and week 4
  The GSRS contains a list of questions on subject's well-being within the period from subject's last visit to study site. The modified Lanza scale is utilized to grade the degree of gastritis
Changes in GSRS as compared to visit 1 (baseline) in each treatment group | Baseline, week 2 and week 4
  The GSRS contains a list of questions on subject's well-being within the period from subject's last visit to study site
Safety assessed by nature, frequency and severity of Adverse Events (AEs) | Up to day 35
  An AE is defined as any untoward medical occurrence in a subject administered a study drug or has undergone study procedures and which does not necessarily have a causal relationship with this treatment
Safety assessed by nature, frequency and severity of Serious Adverse Events (SAEs) | Up to day 35
  Adverse event (AE) is considered "serious" if the investigator or sponsor view any of the following outcomes: Death, life-threatening, persistent or significant disability/incapacity, congenital anomaly or birth defect, hospitalization, or medically important events
Number of participants with Physical Exam abnormalities and/or adverse events related to treatment | Up to day 35
  Number of participants with potentially clinically significant physical exam values
Number of participants with vital signs abnormalities and/or adverse events related to treatment | Up to day 35
  Number of participants with potentially clinically significant vital sign values
Safety assessed through esophagogastroduodenoscopy | Up to day 35
  Amount of gastric content and its nature (mucus, bile, blood), gastric mucosa condition (edema, hyperemia, erosions, mucosal hemorrages, atrophy, hypertrophy) shall be evaluated during esophagogastroduodenoscopy
Number of participants with laboratory value abnormalities and/or adverse events related to treatment | Up to day 35
  Number of participants with potentially clinically significant laboratory values

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Astellas Pharma Russian affiliate
Locations (5):
- Russia (5):
  - Site RU70001, Moscow
  - Site RU70008, Saint Petersburg
  - Site RU70012, Saint Petersburg
  - Site RU70006, Volgograd
  - Site RU70013, Volgograd

IPD SHARING:
Plan to Share IPD: Undecided